CLINICAL TRIAL: NCT05458544
Title: A Phase 1 Open-label, Dose-finding Multi-center Trial of [177Lu]Ludotadipep in Metastatic Castration-resistant Prostate Cancer Patients, Followed by an Open-label, Repeat Dose, Multi-center Phase 2a Trial to Assess Safety and Efficacy
Brief Title: [Lu-177]Ludotadipep in Castration-resistant Prostate Cancer(CRPC): Investigation of Drug and Application
Acronym: LUCIDA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: FutureChem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FC705-US-1
Record Dates: First submitted 2022-06-10; First posted 2022-07-14 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [177Lu]Ludotadipep 3.7 GBq (Experimental): If investigators observed one or no DLT in 6 patients at the 3.7 GBq dose level, the study can advance to the Phase 2a part of the trial after the safety review committee (SRC) review.
  Interventions: Drug: [177Lu]Ludotadipep 3.7 GBq

INTERVENTIONS:
Drug: [177Lu]Ludotadipep 3.7 GBq — Phase 1:
  Patients will receive a single dose of 3.7 GBq of [177Lu]Ludotadipep
  * Test article code/name: [177Lu]Ludotadipep
  * Administration route: intravenous injection
  * Total dose strength: 3.7 GBq
  * Dosage form: solution for injection
  Phase 2a:
  Patients will receive 3.7 GBq of [177Lu]Ludotadipep every 8 [±1] weeks (4 to 6 times)
  * Test article code/name: [177Lu]Ludotadipep
  * Administration route: intravenous injection
  * Total dose strength: 4 to 6 x 3.7 GBq
  * Dosage form: solution for injection

SUMMARY:
Phase 1: The objective of the Phase 1 part of the clinical trial is to verify safety and tolerability (dose-limiting toxicity [DLT], maximum tolerated dose [MTD]) of a single 3.7 Giga-Becquerel (GBq) dose with the potential for one dose level de-escalation to 2.775 GBq if necessary, to determine the recommended [177Lu]Ludotadipep dose for use in the Phase 2a part of the trial.

Phase 2a: The objective of the Phase 2a part of the trial is to evaluate safety and efficacy for repeated administration of the recommended [177Lu]Ludotadipep dose. The Recommended Phase 2 dose (RP2D) will be based on the study results from the Phase 1 trial in South Korea upon consultation with the FDA.

DETAILED DESCRIPTION:
Phase 1:

The patient will attend a Screening visit (-28 to -1 days) prior to study treatment, where it will be determined if the patient is eligible to, and consents to, participate in the trial based on the inclusion/exclusion criteria. [Ga-68]PSMA-11 positron emission tomography (PET)/CT scan will be performed at screening.

Patients who are finally registered for trial participation will be injected with a single dose of [177Lu]Ludotadipep. Ice packs and other cooling therapies will be applied to the major salivary glands from 30 minutes before the administration of [177Lu]Ludotadipep to 60 minutes after the administration to prevent side effects such as sialadenitis. Amino acid solution will be administered slowly intravenously for renal protection over approximately 4 hours from 30 minutes before treatment to 3.5 hours after treatment. 500 mL of 0.9% sodium chloride (NaCl) will be administered slowly intravenously for hydration over approximately 90 minutes from 30 minutes before treatment to 60 minutes after treatment.

Adverse events and DLTs will be assessed continuously for the duration of the 8 [±1] week study period. Other measurements, corresponding to secondary outcomes, are detailed in the Schedule of Assessments and include concomitant medications, laboratory tests, physical examination, vital signs, Eastern cooperative oncology group performance status (ECOG PS), imaging (positron emission tomography-computed tomography [PET/CT], bone scan and Whole Body Scan (WBS)). Follow-up will occur at scheduled visits 1, 2, 4 and 8 weeks after investigational product (IP) administration.

Patients who show a clinical response and who the PI considers will likely benefit from retreatment can be so treated after consultation and agreement of the medical monitor and the sponsor.

Phase 2a:

The patient will attend a Screening visit (-28 to -1 days) prior to treatment with IP, where it will be determined if the patient is eligible to, and consents to, participate in the trial based on the inclusion/exclusion criteria. [Ga-68]PSMA-11 PET/CT and [F-18]FDG-PET scans will be performed at screening.

Patients who are finally registered for trial participation will be injected with a single dose of [177Lu]Ludotadipep. Ice packs and other cooling therapies will be applied to the major salivary glands 30 minutes before and up to 60 minutes after the administration of [177Lu]Ludotadipep to prevent side effects such as sialadenitis. Amino acid solution will be administered slowly intravenously for renal protection over approximately 4 hours from 30 minutes before treatment to 3.5 hours after treatment. 500 mL of 0.9% NaCl will be administered slowly intravenously for hydration over approximately 90 minutes from 30 minutes before treatment to 60 minutes after treatment. WBS or single photon emission computed tomography (SPECT) images will be obtained 24 hours after each administration and Day 7, and AE information will also be captured. Other measurements are detailed in the Schedule of Assessments.

Patients will receive [177Lu]Ludotadipep every 8 [±1] weeks (4 to 6 times).

Patients will be contacted by phone 2 weeks after the first administration for a safety check-up. Four and six weeks after each administration the patient will attend the clinic for a follow-up visit. The following assessments will be performed:

* PSA and other laboratory blood tests (4 and 6 weeks)
* AEs (4 and 6 weeks)
* Urinalysis, physical examination, vital signs, ECOG PS, EORTC QLQ-C30 and Pain Response questionnaires (4 weeks only) The decision on whether to proceed with additional administrations will be determined every 6 weeks after administration of the IP, based on investigator's assessment of tolerability. If a patient does not progress to the next dose administration at 8 weeks, a PSA blood sample will be taken.

A tumor response assessment by CT and bone scan, and additional [Ga-68]PSMA-11 PET/CT and FDG-PET scans will be conducted at end of treatment (EOT). All follow up assessments are detailed in the Schedule of Assessments.

All patients will have long term follow-up every 6 months for 2 years after the last dose of IP unless there is death, withdrawal of consent, or loss to follow-up. Patients who are alive at >2 years after the last dose of IP, unless there is death, withdrawal of consent, or loss to follow-up will be offered participation in a long-term follow-up protocol for up to 10 years. In the long-term survival follow-up, the long-term outcome of the known serious risk of myelosuppression, renal failure, xerostomia, xerophthalmia, and their complications; the potential serious signals of secondary malignancies including myelodysplastic syndrome (MDS), and acute myeloid leukemia (AML); and other serious adverse reactions, will be monitored.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria in order to be included in both the Phase 1 and Phase 2a parts of the trial:

1. Male and ≥ 18 years
2. Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features at initial diagnosis
3. Disease progression on any one of the following: prior enzalutamide, abiraterone, apalutamide or related agent therapy as defined by meeting at least one of the following criteria per the investigator in accordance with the Prostate Cancer Working Group 3 (PCWG3) criteria [Scher et al, 2016]:

   1. PSA progression as defined by a minimum of two rising PSA levels at least 1 week apart, ideally three successive measurements
   2. Soft tissue disease progression defined as >20% increase in sum of diameters of all target lesions based on sum of diameters since treatment started or the appearance of 1 or more new lesions by RECIST 1.1
   3. Bone disease progression defined by two or more new lesions on bone scan
4. Serum testosterone level < 50 ng/dL (< 0.5 ng/mL, < 1.7 nmol/L). Patients may have ongoing androgen deprivation therapy (ADT) with a luteinizing hormone-releasing hormone (LHRH) "super-agonist" or antagonist, and/or be surgically or medically castrated.
5. Patients must have PSMA positive lesions. These are defined as having Ga 68-PSMA-11 uptake greater than that of liver parenchyma in one or more metastatic lesions of any size in any organ system. PSMA-negative lesions are defined as having PSMA uptake equal to or lower than that of liver parenchyma in any lymph node with a short axis of at least 2.5 cm, in any metastatic solid-organ lesions with a short axis of at least 1.0 cm, or in any metastatic bone lesion with a soft-tissue component of at least 1.0 cm in the short axis.
6. Patients receiving bisphosphonate therapy must have been on stable doses for at least 4 weeks prior to Day 1
7. Patients who have received a taxane or are ineligible or choose not to receive taxane-based chemotherapy based on personal preference or physician opinion. Examples of conditions that could make a patient ineligible or refuse to receive taxane-based chemotherapy include the following:

   1. Poor performance status
   2. Prior intolerance to cytotoxic agents
   3. Other serious medical conditions such as symptomatic peripheral neuropathy Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or higher; or clinically significant cardiovascular disease per the Investigator
8. ECOG PS of 0 to 2 for Phase 1 and 0 to 1 for Phase 2a
9. Estimated life expectancy of at least 3 months for Phase 1 and 6 months for Phase 2a as determined by the Investigator.
10. For patients who have partners of childbearing potential, the partner and/or patient must use a method of birth control with adequate barrier protection, deemed acceptable by the principal investigator during the study and for 3 months after last study drug administration.
11. Able and willing to provide signed informed consent and comply with protocol requirements

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria (applies to both Phase 1 and Phase 2a):

1. Impaired organ function as evidenced by the following laboratory values at Screening:

   1. Absolute neutrophil count < 1500/μL
   2. Platelet count < 100,000/μL
   3. Hemoglobin < 9.0 g/dL Note: the patient cannot have received blood transfusion or growth factor support in the 2 weeks prior to screening laboratory hematology assessments.
   4. Albumin < 3.0 g/dL (30 g/L)
   5. Total bilirubin > 2 x upper limit of normal (ULN) unless in instances of known or suspected Gilbert's disease
   6. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN
   7. Calculated creatinine clearance < 60 mL/min (Cockroft-Gault equation), or currently on renal dialysis
2. QT interval corrected for heart rate (QTcF) > 470 msec
3. Sjogren's syndrome
4. Known or suspected brain metastasis or active leptomeningeal disease
5. History of other malignancy within the previous 3 years, except basal cell or squamous cell carcinoma, or non-muscle invasive bladder cancer
6. History of active thromboembolism within the last 3 months of Day 1
7. Serious persistent infection within 14 days prior to Day 1
8. If the patient is known to have a positive polymerase chain reaction (PCR) test for active COVID-19 infection or signs or symptoms consistent with COVID-19, in the absence of a positive PCR test, within 5 days from date of consent
9. Patients with any medical condition or other circumstances that, in the opinion of the investigator, compromise obtaining reliable data, achieving study objectives, or completing the study
10. History of congestive heart failure New York Heart Association (NYHA) class III or IV, uncontrolled hypertension or evidence of coronary artery disease (including a myocardial infarction) within the previous 6 months from date of consent
11. Patients who received any anti-tumor therapy within 4 weeks of Day 1, with the exception of abiraterone, enzalutamide or apalutamide, GnRH therapy and non-radioactive bone-targeted agents
12. Superscan as evidenced on baseline bone scan
13. Treatment with Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 within 6 months prior to Day 1
14. Prior hemi-body irradiation
15. Prior PSMA-targeted radioligand therapy
16. Major surgery within 4 weeks of Day 1
17. Prior systemic beta-emitting bone-seeking radioisotopes
18. Radiation therapy for treatment of prostate cancer within 4 weeks of Day 1
19. Use of anticoagulants within 3 months prior to Day 1 for patients with a history of thromboembolic conditions. Note: Patients receiving anticoagulants for atrial fibrillation are eligible for the study so long as they are on a stable dose of anticoagulants
20. Prior use of any herbal products known to decrease PSA levels (e.g., PC-SPES [prostate cancer hope - dietary supplement] or saw palmetto) within 30 days prior to Day 1
21. Planned initiation of alternative therapy for prostate cancer, investigational therapy, or participation in clinical trials during the study
22. Known history of human immunodeficiency virus (HIV) hepatitis B or C infection:

    1. HIV infected patients who are healthy and have a low risk of Acquired Immune Deficiency Syndrome (AIDS)-related outcomes will be included.
    2. Patients with a history of hepatitis B or C will be allowed to enrol if hepatitis B virus (HBV) DNA or hepatitis C virus (HCV) RNA are undetectable. At this early stage of development, about the main concern is the potential for re-activation or worsening of HBV or HCV from the effect of radiation on lymphocyte function.
23. Vulnerable patients (the investigator involved in the study or his/her family, research staff or students of the investigator involved in the study)
24. Implantation of investigational medical device within 4 weeks of Day 1 or current enrolment in oncologic investigational drug or device study
25. Use of investigational drugs within 4 weeks or less than 5 half-lives of Day 1
26. Patients are excluded if treatment other than the treatment provided in this study is determined more appropriate as determined by the investigator based on the patient and disease characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and ≥ 18 years
Enrollment: 26 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) with a single fixed dose of [177Lu]Ludotadipep during the first cycle (8 [±1] weeks) (Phase 1) | Single dose and 8 weeks follow up (Screening up to 28 days)
  Determination of Maximum Tolerated Dose (MTD)
Objective Response Rate (Phase 2a) | up to 40 weeks (4 to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  Complete Response [CR] Rate + Partial Response [PR] Rate

SECONDARY OUTCOMES:
Safety assessments (Phase 1) | Single dose and 8 weeks follow up (Screening up to 28 days)
  Safety assessments will include the recording of AEs from the time of signing the informed consent form (ICF), laboratory tests, electrocardiograph (ECG), vital signs, physical examinations and Eastern Cooperative Oncology Group Performance Status (ECOG PS).
Whole-body absorbed dose (Phase 1) | Single dose and 8 weeks follow up (Screening up to 28 days)
  Whole-body absorbed dose of [177Lu]Ludotadipep biodistribution parameters will be performed as follows:
  1. Analysis will be conducted on data collected approximately 2 hours, 24 hours, 48 hours and 7 days after injection with IP using the obtained WBS images.
  2. Aspects on biodistribution will be confirmed in WBS images.
  3. A chart will be prepared with confirmed values for each organ, and a descriptive and comparative analysis will be conducted for the changes over time.
Biodistribution: assessment of the absorption (uptake) into the blood, lungs, liver, spleen, pancreas, kidneys, muscle, stomach, and tumor based on the level obtained from whole body scan (WBS) 2 hours, 24 hours, 48 hours, and 7 days post-dose (Phase 1) | Single dose and 8 weeks follow up (Screening up to 28 days)
  The assessment of [177Lu]Ludotadipep biodistribution parameters will be performed as follows:
  1. Analysis will be conducted on data collected approximately 2 hours, 24 hours, 48 hours and 7 days after injection with IP using the obtained WBS images.
  2. Aspects on biodistribution will be confirmed in WBS images.
  3. A chart will be prepared with confirmed values for each organ, and a descriptive and comparative analysis will be conducted for the changes over time.
Disease Control Rate (Phase 2a) | up to 40 weeks (4 to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  Disease Control Rate (DCR) = Complete Response Rate (CR) + Partial Response Rate (PR) + Stable Disease Rate (SD)
Safety assessments (Phase 2a) | up to 40 weeks (4 to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  Safety assessments will include the recording of Adverse event (AEs) from the time of signing the Informed consent form (ICF), laboratory tests, Electrocardiograph (ECG), vital signs, physical examinations and Eastern cooperative oncology group performance status (ECOG PS).
Prostate Specific Antigen Response Rate (PSA RR) (Phase 2a) | up to 40 weeks (4 to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  Defined as the proportion of participants with a PSA reduction of ≥ 50% from baseline
Tumor response rate (Phase 2a) | up to 40 weeks (4 to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  Defined as the proportion of participants with a confirmed CR or PR divided by the total number of participants (using Response Evaluation Criteria in Solid Tumors 1.1 [RECIST 1.1])
Pain response rate (Phase 2a) | up to 40 weeks (4 to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  Defined as: ≥2 point reduction in Present Pain Intensity Scale (PPI) score from baseline with no increase in analgesic score; and/or ≥50% decrease in analgesic score with no increase in PPI using the Short Form McGill Questionnaire (SF-MPQ)
European Organization for Research and Treatment of Cancer quality of life (EORTC QLQ-C30) questionnaire (Phase 2a) | up to 40 weeks (4 to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients.
Time to death for any reason (Overall Survival [OS]) (Phase 2a) | up to 40 weeks (4 to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  Defined as time from initiation to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Arif Hussain, MD, Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - VA Greater Los Angeles Healthcare System,Cancer Center Research, Los Angeles, California
  - University of Maryland, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Pennsylvania Cancer Specialists & Research Institute (Formerly Gettysburg Cancer Center), Gettysburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No